

## A Randomized, Phase II, Open-Label Study Evaluating the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients with Chronic Pain, Anxiety, Depression, and/or Sleeplessness

PROTOCOL NUMBER: Nu-V3P2RCT

PROTOCOL NAME: Nu-V3 RCT Protocol

**INVESTIGATIONAL PHASE:** Phase II

VERSION: 1.6

NCT NUMBER: NCT05335980

**INVESTIGATIONAL DEVICE**: Nu-V3

ORIGINAL PROTOCOL ISSUE DATE: April 20, 2022

**VERSION DATE:** April 20, 2022

**STUDY SPONSOR:** Nu-Life Solutions

5252 E 82nd St., Suite 200 Indianapolis, IN 46250

**United States** 

#### **STUDY CONTACTS:**

Medical MonitorClinical Trial ManagerBiostatisticianVipul Kella, MDEric T. SiebeneckJason Sutherlandvkella@nu-(317)941-6709jsutherland@nu-lifesolutions.comlifesolutions.com

#### **CONFIDENTIALITY STATEMENT**

This document is the property of Nu-Life Solutions. It contains confidential and proprietary information belonging to Nu-Life Solutions; therefore, its use is intended solely for physicians, clinical research staff, and contract research organizations ("study personnel") participating in clinical studies of Nu-V3. Reproduction is authorized for and strictly limited to study personnel for Nu-Life Solutions, reproduction for any other purpose is prohibited.

#### **Sponsor Protocol Signature:**

## **Protocol Signature Page**

# A Randomized, Phase II, Open-Label Study Evaluating Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients with Chronic Pain, Anxiety, Depression, and/or Sleeplessness

Protocol Amendment 1.6: April 20, 2022

By signing below, the Investigator attests that they will adhere to the protocol and Informed Consent Form and report, to the Study Sponsor and the IRB, any adverse device or participant study event.

| Investigator Name: |
|--------------------|
| Title: |
| Address: |
| Address: |
| Address: |
| Phone: |
| Facsimile: |
| Signature: |
| Date: |

## Table of Contents

| 1.0 Introduction | 4 |
|-----------------------------------------------------------|----|
| 1.1 Background | 4 |
| 1.2 Device Description | 5 |
| 1.3 Non-significant Risk Medical Device Study | 6 |
| 2.0 STUDY OBJECTIVE | 6 |
| 3.0 STUDY PARTICIPANT SELECTION CRITERIA | 6 |
| 3.1 Inclusion Criteria | 6 |
| 3.2 Exclusion Criteria | 6 |
| 4.0 STUDY PROTOCOL | 7 |
| 4.1 Phase II Study Assessment Tables | 9 |
| 5.0 DATA COLLECTION AND RETENTION | 11 |
| 6.0 DATA DISCLOSURE AND SUBJECT CONFIDENTIALITY | 11 |
| 7.0 ADVERSE EVENT(S) | 11 |
| 8.0 STUDY ENDPOINT and DATA ANALYSIS | 12 |
| 8.1 Primary Endpoints | 12 |
| 8.2 Secondary Endpoints | 13 |
| 8.3 Sub-Analyses | 14 |
| 9.0 STUDY MONITORING | 14 |
| 10.0 REFERENCES CITED | 15 |
| Appendix 1: STUDY PROCESS MAPS | 17 |
| Appendix 2: ELIGIBILITY CHECKLIST | 18 |
| Appendix 3: IRB UNANTICIPATED PROBLEM FORM | 20 |
| Appendix 4: ADVERSE EVENT FORM | 22 |
| Appendix 5: MEDICAL HISTORY FORM | 23 |
| Appendix 6: TREATMENT FORM | 27 |
| Appendix 7: MEDICATIONS FORM | 28 |
| Appendix 8: EPRO QUESTIONNAIRES | 30 |
| Appendix 9: Baseline Symptom Quetionnaire for Eligibility | 38 |

#### 1.0 Introduction

## 1.1 Background

Research evidence has shown that the symptoms of chronic pain, anxiety, depression, and sleeplessness, or any combination of these symptoms are prevalent among patient populations with chronic medical conditions, particularly inflammatory arthritis (Psoriatic Arthritis, Rheumatoid Arthritis), Fibromyalgia, anxiety disorders (PTSD, Generalized Anxiety Disorder), Depression, Chronic Pain conditions (neuropathy, chronic neck and back pain, Osteoarthritis, TMJ Syndrome), and sleep disorders. Patients with one of these chronic conditions often have clusters of one or more of these four symptoms (pain, anxiety, depression, and/or sleeplessness).

These patient populations have a need for an innovative treatment approach to address these symptoms, as they often occur simultaneously. By addressing all possible combinations of these symptoms in an individual patient or population, significant improvements in patients' health and health outcomes can be achieved.

Globally, the lifetime prevalence of anxiety disorders from a 2013 meta-analysis was 7.3% (4.8-10.9%) and ranged from 5.3% (3.5-8.1%) in African cultures to 10.4% (7.0-15.5%) in Euro/Anglo cultures.<sup>1</sup> These statistics translate into 1 out of 13, and 1 out of 10 people affected globally and in North America, respectively. In the United States alone, anxiety affects about 18% of the population or 40 million adults aged 18 and older at cost of more than \$42 billion a year in 1990.<sup>2,3</sup>

In a separate systematic review on depression, the global prevalence of major depressive disorder was 4.7% (4.4-5.0%).<sup>4</sup> In 2015, over 16 million adults aged 18 or older have been estimated to have had at least one major depressive episode in the prior year, representing 6.7% of all U.S. adults.<sup>5</sup>

Insomnia is a global public health issue and is believed to affect approximately 30-35% of the global population.<sup>6,7</sup> Poor sleep has been associated with decreased immunity, depression, anxiety, poorer quality of life, obesity, increased pain, occupational errors, absenteeism from work, and motor vehicle crashes.<sup>7,8</sup>

The prevalence of chronic pain, like all the previous conditions discussed, is highly variable among subgroups in population and by indication. It is estimated that approximately 20% of the adult European population suffers from chronic pain. Similarly, approximately 17.6% (about 40 million) of US adults experience severe levels of pain along with over 11.2% (25.3 million) of adults suffering from daily pain for the prior 3 months at an annual estimated cost of approximately \$560-\$635 billion. 10,11

Given the high prevalence of conditions associated with chronic pain, anxiety, depression, and/or sleeplessness (CPADS), the associated economic burden, and lack of safe and cost-effective therapies, interest and research is expanding into the field of neuromodulation therapies, including TENS devices, to meet this need.

The Nu-V3 device is not considered to be a Transcutaneous Electrical Nerve Stimulation (TENS) device. TENS devices are applied only in the area of the body directly related to the pain. The Nu-V3 device is placed on the auricular (ear) area and utilizes a non-invasive electrical micro-signal to access the cranial nerves via three small electro-gel pads. There are no TENS devices currently approved or cleared by the FDA that qualify as being substantially equivalent.

Under further research pertaining to accessing the cranial nerves, in particular the vagus nerve, we discovered that there are a variety of Vagal Nerve Stimulators available. However, none are non-invasive and small enough to be attached to the ear while stimulating multiple cranial nerves in the auricular area.

In summary, while Nu-V3 is technically a transcutaneous device, the mechanism for mitigation of symptoms (chronic pain, anxiety, depression, and sleeplessness) is unique by TENS standards for the following reasons:

- A. TENS is typically placed in the general area where the pain exists. Nu-V3 is placed only in the auricular area (on the ear) and accesses the cranial nerves as the mechanism for relief.
- B. TENS devices are known to stimulate muscular tissue and nerves in the area where pain exists, creating vasodilation (increased blood flow) and thereby the possibility of temporary relief. Nu-V3, by accessing the cranial nerves (specifically the vagus nerve) non-invasively, acts to stimulate the body's natural enkephalins and elevate blood flow, and may result in the balancing or rebalancing of the Autonomic Nervous System (ANS).<sup>12-18</sup>
- C. By accessing the cranial nerves in the manner described above, the effect may be cumulative and residual and offer the patient immediate, intermediate, and longer lasting relief from their symptoms.

In part, the purpose of this clinical study is to demonstrate the effect of the device upon the four specific symptoms of chronic pain, anxiety, depression, and sleeplessness. Any one or combination of these symptoms may result in Autonomic Nervous System dysfunction.

## 1.2 Device Description

The Nu-V3 device is a miniaturized, wearable, microchip-controlled, cranial nerve stimulation treatment device which delivers pulsed micro-signals over a period of 14 days. The Nu-V3 device provides a continuous flow of intermittent, low frequency electrical pulses to the ear's specific cranial nerve endings. The Nu-V3 device is a patent pended, non-invasive transcutaneous stimulating device which offers useful features to the patient and clinical professional. The Nu-V3 device control features are set by the manufacturer and prevent patient misuse of the device.

Three miniature, non-invasive, electro-gel pads are utilized to deliver a micro signal at 1

Hz in a square plus minus waveform, which cycles on and off every three hours to provide a resting period and prevent adaption to the stimulation. The device is powered by three (No.10) zinc air batteries at 1.4 volts each (4.2 volts in total), to provide the required stimulation for up to 14 days. The low frequency, reliability of the zinc air batteries and consistency of the micro-signal through the eight-pin micro-chip technology, provides consistent and equivalent stimulation energy regardless of individual skin impedance.

#### 1.3 Non-significant Risk Medical Device Study

The FDA considers other microcurrent transcutaneous devices (such as TENS devices) as nonsignificant risk devices for medical device studies.<sup>19</sup> The Nu-V3 device used in this study reflects an investigational device that meets the definition of a nonsignificant risk device per review of the IRB.

#### 2.0 STUDY OBJECTIVE

The objective of this research study is to collect data which demonstrates the ability of the Nu-V3 device to offer relief from one or more of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness.

## 3.0 STUDY PARTICIPANT SELECTION CRITERIA

#### 3.1 Inclusion Criteria

- Participant is at least 18 years of age
- Participant presents with one or more of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness
- Participants must score greater than or equal to a 5/10 for their primary symptom score on the Baseline Symptom Questionnaire
- Patient's chosen primary symptom must have an available accrual slot for the participant. If patient scores greater than or equal to a 5/10 for a second symptom, they can be selected to accrue to another symptom slot.
- Participant has signed the Informed Consent Form

#### 3.2 Exclusion Criteria

- Participants with a hearing aid
- Participants with a pacemaker
- Participants with irregular heart rate or a heart rate lower than 60 beats per minute (bradycardia)
- Have had a transplant within the last 2 years
- Have had a heart attack or cardiac bypass surgery within the last 12 months
- Patients with complaints of dizziness or lightheadedness within the last 3 months
- Women who are pregnant

- Participants with Diabetic Retinopathy
- Current ear infection
- SBP < 100 and/or DBP < 60</li>
- History of uncontrolled bipolar disorder within the last 12 months
- History of uncontrolled seizures within the last 12 months
- History of aneurysms
- History of syncope within the last 12 months
- Participants that have had a TIA or stroke within the last 12 months
- Participants with health problems deemed at risk for the study by the Principal Investigator
- Participants with any changes to Pain/Anxiety/Depression/Sleeplessness medications within last 60 days (participants that do not meet this medicationchange washout period may be delayed until 60-day period is met)
- Participants that are currently under adjudication process for disability support,
   VA or other

#### 4.0 STUDY PROTOCOL

The Nu-V3 Clinical Study is a randomized, open-label study using the Nu-V3 cranial nerve stimulation treatment device in patients with chronic pain, anxiety, depression, and/or sleeplessness. Study participants are those who have signed the informed consent form, met the inclusion and exclusion criteria, and are enrolled in the study at one of multiple sites.

Subjects randomized to receive the Nu-V3 treatment will undergo the following regimen:

- At the baseline visit, patients will be asked to complete study questionnaires (Appendix 11) regarding all of the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their quality of life, active medications, medical history, and demographical information. The subject's primary symptom of concern will also be notated at baseline, for later assessment of continuation after week 12.
- At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their activity level and quality of life.
- The sessions will begin with the Nu-V3 device being clipped on the ear and three small pads (non-invasive) adhered to the surface of the ear. Each Nu-V3 device lasts for up to 28 days with a change in the pads approximately 7 days into the treatment.
- Each session takes approximately 15-20 minutes. The placement of the device takes approximately 5 minutes, and the remaining time is spent verifying ePRO form completion, and evaluating the patient for all device effects.
- The Nu-V3 device is mobile and is worn externally on the left ear 24 hours a day during treatment, fitting comfortably behind the ear. An electrical signal is sent to

- the external ear through coated wire leads attached to the device and adhesive pads which attach to three sites on the ear.
- Participants should be able to perform their typical day-to-day activities while wearing the device. They may shower while wearing the Nu-V3 device, if they do not get the device wet and use the small disposable ear covers that are provided for them.
- In the event the Nu-V3 gel pads are inadvertently removed or the device comes
  off, the participant will contact the site coordinator. The participant is
  encouraged to adjust the device placement as needed for comfort.
- Patients should not change their existing forms of treatment or medications without discussion with the study investigator.

Subjects randomized to the observation control arm of the study will undergo the following regimen:

- At the baseline visit, patients will be asked to complete study questionnaires (Appendix 11) regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their quality of life, active medications, medical history, and demographical information. The subject's primary symptom of concern will also be notated at baseline.
- At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: chronic pain, anxiety, depression, and/or sleeplessness, as well as their activity level and quality of life.
- Patients should not change their existing forms of treatment or medications without discussion with the study investigator.
- At completion of 12 weeks of standard of care treatment post study enrollment, observation (control arm) subjects will be offered a crossover into the treatment arm of the study for an additional 24 weeks.

#### Sample size

For this Phase II study, a total of 100-200 subjects will be randomized 1:1 to either the Nu-V3 treatment arm or to the observation treatment arm (SOC, control).

#### Recruitment

Participants are enrolled into relevant symptom cohorts based on their chronic pain, anxiety, depression, and/or sleeplessness symptom presentation at baseline and treated with the Nu-V3 device for 24 weeks.

#### Analyses

Interim analysis of reported data will be based on baseline symptom cohort and conducted at 6, 12, 18, and 24 weeks during this time. The participant will be evaluated after the initial 12-week treatment period to assess for further therapeutic need. Upon having three consecutive weeks of mean symptom reduction of ≥70% via patient reported numerical scales, the participant will continue as described in the study assessments table, but without device therapy. Then if the participant's primary

symptom score increases at any time by ≥20%, they may again continue device therapy until week 24, as depicted in section 4.1.

Study subjects randomized to the observation arm will be offered the opportunity to cross-over to the Nu-V3 study treatment arm upon completion of the initial 12-week observation study period.

## 4.1 Phase II Study Assessment Tables

| Nu-Life Solutio | ns<br>Nu] | | Initial Study Assessments Table *Evaluations are completed weekly, every 7 days ±3 days | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nu-V3 Treatment Arm<br>Evaluation* | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5 | Week<br>6 | Week<br>7 | Week<br>8 | Week<br>9 | Week<br>10 | Week<br>11 | Week<br>12 |
| Informed Consent | Х | | | | | | | | | | | |
| Inclusion and Exclusion <sup>1</sup> | х | | | | | | | | | | | |
| Patient Registration <sup>1</sup> | х | | | | | | | | | | | |
| Medications Form <sup>1</sup> | x | | | x | | | | х | | | | х |
| Patient Onboarding and<br>Orientation <sup>2</sup> | х | | | | | | | | | | | |
| In office assessment | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| New Device Placed <sup>3</sup> | х | | | | Х | | | | Х | | | |
| Pad Replaced <sup>3</sup> | | х | х | х | | х | х | х | | х | х | х |
| Treatment Forms <sup>1</sup> | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| No Device | | | | | | | | | | | | |
| HRV Assessment (optional) <sup>4</sup> | x | х | х | x | х | х | х | х | х | х | х | х |
| ePRO Questionnaires <sup>5</sup> | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Patients' Global Impression of Change ePRO form (PGIC) <sup>5</sup> | | х | х | х | х | х | х | х | х | х | х | х |
| Providers' Global Impression of Change ePRO form (PGIC) <sup>1</sup> | | х | | х | | х | | х | | х | | х |
| Optional Patient Media<br>Testimony <sup>6</sup> | х | х | | х | | | | х | | | | х |

- 1. Inclusion/Exclusion, Registration, Medications, Treatment, and Providers' PGIC forms to be completed by site via online module.
- 2. Patient Onboarding and Orientation includes introductory demographics form, Nu-V3 patient training video
- 3. Upon having three consecutive weeks of primary symptom reduction of ≥70% via patient reported numerical scales from baseline, the participant will have reached symptom response plateau and will continue as described in the study assessments table, but without device therapy. Then if the participant's primary symptom score increases at any time by ≥20% from the symptom response plateau, they may again continue device therapy until week 24.
- 4. (Optional) HRV assessment will be conducted before the first treatment and again 15-20 minutes following the first treatment. The HRV assessment will also be conducted prior to each weekly treatment. This assessment is applicable to participating sites per the clinical trial agreement. Contact the clinical trial manager for Information.
- 5. ePRO questionnaires completed on patient's mobile device: DQ-9 (baseline), PTB-7, PEG, GAD-7, PHQ-9, PROMIS 4a, PGIC
- 6. If patient consents to media testimony, site will collect via study collection process.

| Nu-Life Solutio | Study Assessments Table *Evaluations are completed weekly, every 7 days ±3 days | | | | | | | | | Nu-V³ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nu-V3 Treatment Arm<br>Evaluation* | Week<br>13 | Week<br>14 | Week<br>15 | Week<br>16 | Week<br>17 | Week<br>18 | Week<br>19 | Week<br>20 | Week<br>21 | Week<br>22 | Week<br>23 | Week<br>24 |
| Medications Form <sup>1</sup> | | | | х | | | | х | | | | х |
| In office assessment | х | х | | х | х | | х | х | | х | х | х |
| New Device Placed <sup>2</sup> | х | | | х | | | х | | | х | | |
| Pad Replaced <sup>2</sup> | | х | | | х | | | х | | | х | |
| Treatment Forms <sup>1</sup> | х | х | | х | х | | х | х | | х | х | |
| No Device | | | х | | | х | | | х | | | х |
| HRV Assessment (optional) <sup>3</sup> | х | х | | х | х | | х | х | | х | х | |
| ePRO Questionnaires <sup>4</sup> | х | х | х | х | х | х | х | х | x | х | х | х |
| Patients' Global Impression of Change ePRO form (PGIC) <sup>4</sup> | х | х | х | х | х | х | х | х | х | х | х | х |
| Providers' Global Impression of Change ePRO form (PGIC) <sup>1</sup> | | х | | | х | | | х | | х | х | |
| Optional Patient Media<br>Testimony <sup>5</sup> | х | х | | х | | | · | х | · | · | | х |

- 1. Providers' PGIC form, Medications and Treatment forms to be completed by site via online module.
- Upon having three consecutive weeks of mean symptom reduction of ≥70% via patient reported numerical scales, the participant will
  continue as described in the study assessments table, but without device therapy. Then if the participant's primary symptom score
  increases at any time by ≥20%, they may again continue device therapy until week 24.
- 3. (Optional) HRV assessment before the first treatment and again 15-20 minutes following the first treatment. HRV assessment will also be conducted prior to each weekly treatment. This assessment is applicable to participating sites per the clinical trial agreement. Contact the clinical trial manager for Information.
- 4. ePRO questionnaires completed on patient's mobile device: DQ-9 (baseline), PTB-7, PEG, GAD-7, PHQ-9, PROMIS 4a, PGIC
- 5. If patient consents to media testimony, site will collect via study collection process.

| Nu-Life Solution | Control Study Assessments Table *Evaluations are completed weekly, every 7 days ±3 days | | | | | | | | | Nu-73° | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Control Arm<br>Evaluation* | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5 | Week<br>6 | Week<br>7 | Week<br>8 | Week<br>9 | Week<br>10 | Week<br>11 | Week<br>12 |
| Informed Consent | х | | | | | | | | | | | |
| Inclusion and Exclusion <sup>1</sup> | x | | | | | | | | | | | |
| Patient Registration <sup>1</sup> | х | | | | | | | | | | | |
| Medications Form <sup>1</sup> | х | | | х | | | | х | | | | х |
| Patient Onboarding and<br>Orientation <sup>2</sup> | х | | | | | | | | | | | |
| In office assessment | х | | | х | | | | х | | | | х |
| No Device | х | х | х | х | х | х | х | х | Х | х | х | х |
| ePRO Questionnaires <sup>3</sup> | х | | | х | | | | х | | | | х |
| Patients' Global Impression of Change ePRO form (PGIC) <sup>3</sup> | | | | х | | | | х | | | | х |

- 1. Inclusion/Exclusion, Registration, Medications, Treatment, and Providers' PGIC forms to be completed by site via online module.
- 2. Patient Onboarding and Orientation includes introductory demographics form, Nu-V3 patient training video
- 3. ePRO questionnaires completed on patient's mobile device: DQ-9 (baseline), PTB-7, PEG, GAD-7, PHQ-9, PROMIS 4a, PGIC

#### 5.0 DATA COLLECTION AND RETENTION

The study endpoints data will be collected from each participant's study questionnaires. The data will be collected electronically via the patient's own device and uploaded to an electronic data capture system. The data will be used to measure whether the Nu-V3 device provides participants with a reduction in participants' chronic pain, anxiety, depression, and/or sleeplessness.

The data analysis will include baseline data for each participant's questionnaire prior to beginning treatment with the Nu-V3 device. Longitudinal data will consist of participant's weekly questionnaires measuring chronic pain, anxiety, depression, and sleeplessness during the treatment phase. The final data collection will be completed by participants at the end of the treatment with the Nu-V3 device and will measure chronic pain, anxiety, depression, and sleeplessness.

The Principal Investigator at each site will be responsible for recording, collecting, and storing the research participant's study data. The written records will be stored in a secure location. Only the Principal Investigator or designated study staff will have access to the study records and all electronic files will be password protected. The Principal Investigator will also maintain adequate records for the study including:

- all correspondence with the IRB and Sponsor
- other pertinent data related to the study

All records are to be retained by the Principal Investigator for a period of three (3) years following the closure of the study. Following study closure, the Principal Investigator shall inform Nu-Life of the location of study records and storage changes (i.e., the Principal Investigator leaves the institution where the study was conducted). In such cases, the study records may be transferred to another institution, investigator, or to Nu-Life upon written agreement between the Principal Investigator and Nu-Life.

#### 6.0 DATA DISCLOSURE AND SUBJECT CONFIDENTIALITY

Medical record confidentiality and data protection will be maintained at every visit. Subject medical information obtained because of this study is considered confidential and disclosure to third parties, other than those noted below, is prohibited. Data generated during this study is to be available for inspection on request by the FDA or other government regulatory agency auditors, the Sponsor's authorized representatives, and the IRB.

## 7.0 ADVERSE EVENT(S)

Subjects will be evaluated for safety if they have received any study treatment. Adverse event assessments will be continuous during the 24-week trial (see section 4.1). During

treatment visits, toxicity assessments should be done in person. Once subjects reach symptom stabilization and are not actively receiving device therapy, follow-up either in person or documented via telephone call, is acceptable. Adverse events and will be graded according to the NIH-CTCAE version 5.0.

Potential unanticipated problems require prompt reporting to the central IRB and study sponsor. These problems potentially place subjects or others at greater risk of physical or psychological harm than was previously recognized, and warrant consideration of substantive changes in the protocol or informed consent process or other action to protect the safety, welfare, or rights of participants. The central IRB must be notified within 5 calendar days of the event and the study sponsor within 24 hours. The completed IRB Unanticipated Problem Form (Appendix 7) must be received by the central IRB within 10 calendar days of the event to avoid a major deviation.

Unanticipated problems are defined as those problems which alter the risks to subjects or others. This includes any study suspensions or holds. This form will be used to report any problem that is unforeseen or involves risk. One form will be used per event or problem.

#### 8.0 STUDY ENDPOINT and DATA ANALYSIS

8.1 Primary Endpoints: Primary endpoints consisted of the following:

<u>Safety</u>: At screening/baseline, a medical history will be obtained to capture relevant underlying conditions. The screening/baseline examinations will include BP, and HR. Baseline signs and symptoms are those that are assessed within 14 days prior to week 1 treatment.

Concomitant medications will be collected from within 14 days prior to enrollment through the study treatment period and maintenance period (see Study Assessments Table section 4.1).

The primary safety endpoint is the occurrence of reported unanticipated problems involving risk to subjects or others ("UPIRTSOs"). These UPIRTSOs are defined as those problems which alter the risks to subjects or others. This includes any study suspensions or holds. The primary safety endpoint analyses will be based on a risk-benefit conclusion.

<u>Effectiveness</u>: There are four instruments measuring participant's symptoms of chronic pain, anxiety, depression, and sleeplessness. The primary effectiveness endpoint is a statistically significant reduction in one or more of measures of: chronic pain, anxiety, depression, or sleeplessness between baseline and 12 or 24 weeks after initiating treatment.

The null hypothesis to disprove is that there is no statistically significant reduction from baseline to 12 or 24 weeks in mean chronic pain, anxiety,

depression, or sleeplessness symptom severity scores using the Nu-V3 device compared with the usual care cohort.

The instruments used in this study are:

Chronic Pain – Pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G) (PEG Scale),

The PEG is a three-item instrument that measures pain intensity (one item) and pain interference (two items). Each item is valued from 0 (no pain/interference) to 10 (as bad as you can imagine). The instrument score is calculated as the average of the three item values.

Anxiety - Generalized Anxiety Disorder 7-item (GAD-7)

The GAD-7 is a seven-item instrument that measures respondents' symptoms of anxiety. Each item is scored on a four-point Likert scale, and values range from 0 ("Not at all") to 3 ("Nearly every day".) Items are summed to determine the instrument's score. Values of 10 or higher have been associated with moderate anxiety, while values of 15 or higher have been associated with severe anxiety.

Depression - Patient Health Questionnaire (PHQ-9)

The PHQ-9 is a nine-item instrument that measures depression-related symptoms and functional impairment. Each item is scored on a four-point Likert scale and values range from 0 ("Not bothered at all") to 3 ("Bothered nearly every day.") The items' values are summed to determine the instrument's score. PHQ-9 values of 10 and 15 represent moderate and moderately severe depression respectively.

Sleeplessness - PROMIS short form 4a

This eight item instrument measures sleep disturbance and sleep-related impairment.

## 8.2 Secondary Endpoints: Secondary endpoints consisted of the following:

<u>Effectiveness:</u> There are two secondary effectiveness endpoints:

- 1. In the Nu-V3 device treatment arm, the study will report the mean time from treatment initiation to reduction of symptoms of at least 30% in any of the four domains of symptom measurement.
- 2. In both the Nu-V3 device treatment arm and the observation arm, the study will report the mean percentage change in symptoms severity from initiation to 12 and 24 weeks for each instrument.

Additional secondary endpoints of this study are:

 Mean improvement in quality of life measured with Patient's Global Impression of Change (PGIC) between the treatment and usual care arm, and

• Mean improvement in activities of daily living via Perceived Treatment Benefit Form (PTB-6) between the treatment and usual care arm.

#### 8.3 Sub-Analyses: Sub-Analyses consist of the following:

The study has several sub-analyses. They include:

- The mean number of weeks that chronic pain, anxiety, depression, and sleeplessness response are achieved and sustained, without utilization of another device or change in other treatments, during the full 24-week intervention in the Nu-V3 device treatment arm.
- The mean number of weeks to initial benefit from Nu-V3 device use in the Nu-V3 device treatment arm. Benefit is defined as a reduction of at least 30% of symptoms in at least one of chronic pain, anxiety, depression, or sleeplessness.
- The device's comfort-of-use, and patient's perceived treatment benefit in the Nu-V3 device treatment arm.

#### 9.0 STUDY MONITORING

Nu-Life will monitor the study according to good clinical practice. Monitoring will begin upon enrollment of the first 5 patients at the site and will continue every 8 weeks until completion of the study. The Principal Investigator will work with a representative from Nu-Life to ensure the study is conducted according to this protocol and that all study matters are properly communicated.

#### **10.0 REFERENCES CITED**

- 1. Baxter AJ, Scott KM, Vos T, Whiteford HA. <u>Global prevalence of anxiety disorders: a systematic review and meta-regression.</u> Psychol Med. 2013 May;43(5):897-910.
- 2. *National Institutes of Health*. U.S. Department of Health and Human Services, n.d. Web. 25 Jan. 2017.
- 3. Greenberg PE, Sisitsky T, Kessler RC, et al. <u>The economic burden of anxiety disorders in the 1990s.</u> J Clin Psychiatry. 1999 Jul;60(7):427-35.
- 4. Ferrari, A.J., Somerville, A.J., Baxter, A.J., Norman, R., Patten, S.B., Vos, T. and Whiteford, H.A. (2013) 'Global variation in the prevalence and incidence of major depressive disorder: a systematic review of the epidemiological literature', *Psychological Medicine*, 43(3), pp. 471–481.
- 5. Center for Behavioral Health Statistics and Quality. (2016). Key substance use and mental health indicators in the United States: Results from the 2015 National Survey on Drug Use and Health (HHS Publication No. SMA 16-4984, NSDUH Series H-51). Retrieved from http://www.samhsa.gov/data/
- 6. PharmaPoint: Insomnia Global Drug Forecast and Market Analysis to 2023. Feb-2015
- 7. Roth T. Insomnia: Definition, Prevalence, Etiology, and Consequences. *Journal of Clinical Sleep Medicine: JCSM: official publication of the American Academy of Sleep Medicine.* 2007;3(5 Suppl):S7-S10.
- 8. Mai E, Buysse DJ. Insomnia: Prevalence, Impact, Pathogenesis, Differential Diagnosis, and Evaluation. *Sleep medicine clinics*. 2008;3(2):167-174.
- 9. Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333.
- 10. Nahin RL. <u>Estimates of pain prevalence and severity in adults: United States, 2012.</u> *Journal of Pain.* 2015;16(8):769-780.
- "2 Pain as a Public Health Challenge." Institute of Medicine. 2011. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington, DC: The National Academies Press
- 12. Ueno N et al. Innervation of the external ear in humans and musk shrew. Nihon Jibiinkoka Gakkao Kaiho. 1993 Feb;92(2):212-8. Japanese
- 13. He W, Wang X, Shi H, et al. Auricular Acupuncture and Vagal Regulation. Evidence-based Complementary and Alternative Medicine: eCAM. 2012;2012:786839. doi:10.1155/2012/786839
- 14. Jean-Pierre Barral and Alain Croibier, Chapter 25 Ear, In Manual Therapy for the Cranial Nerves, Churchill Livingstone, Edinburgh, 2009, Pages 227-238, ISBN 9780702031007, https://doi.org/10.1016/B978-0-7020-3100-7.50028-8.
- 15. Torsten Liem, Chapter 17 The organ of hearing and balance, In Cranial Osteopathy (Second Edition), Churchill Livingstone, Edinburgh, 2004, Pages 605-633, ISBN 9780443074998, https://doi.org/10.1016/B978-044307499-8.50024-7.
- Terry Oleson, 2 Theoretical Perspectives of Auriculotherapy, In Auriculotherapy Manual (Fourth Edition), Churchill Livingstone, Saint Louis, 2014, Pages 25-86, ISBN 9780702035722, https://doi.org/10.1016/B978-0-7020-3572-2.00002-1.

- 17. Review of the Uses of Vagal Nerve Stimulation in Chronic Pain Management. Chakravarthy K, Chaudhry H, Williams K, Christo PJ. Curr Pain Headache Rep. 2015 Dec;19(12):54. doi: 10.1007/s11916-015-0528-6. Review.
- 18. Pavlov VA, Tracey KJ. The vagus nerve and the inflammatory reflex—linking immunity and metabolism. Nature reviews Endocrinology. 2012;8(12):743-754. doi:10.1038/nrendo.2012.189.
- 19. Information Sheet Guidance for IRBs, Clinical Investigators, and Sponsors,: U.S. Department of Health and Human Services, Food and Drug Administration, Center for Devices and Radiological Health (CDRH), January 2006, http://www.fda.gov/downloads/Regulatory Information/Guidances/UCM126418.pdf

## **Appendix 1: Study Process Maps**

Figure 1- Baseline Visit



Figure 2- Weekly Visits



## **Appendix 2: Eligibility Checklist**



Nu-V3 RCT PROTOCOL

#### SCREENING AND ELIGIBILITY CHECKLIST

| | | SCREENING AND ELIGIBILITY CHECKLIST |
|---|---|---|
| A Rand | A Randomized, Phase II, Open-Label Study Evaluating the Nu-V3 Cranial Nerve Stimulation Treatmen<br>Device in Patients with Chronic Pain, Anxiety, Depression, and/or Sleeplessness | |
| Subject | | |
| | | ation Number: |
| Date of | Consent: | |
| | | OF ELIGIBILITY: □eligible / □ineligible for participation in the study. |
| Investi | gator Sig | nature:Date: |
| Printed | l Name: | |
| answe | ered No | RITERIA (all questions should be answered YES – If question is<br>o, subject is not eligible for participation) |
| Yes | No | |
| | | Participant is at least 18 years of age |
| | | Participant presents with one or more of the following symptoms:<br>chronic pain, anxiety, depression, and/or sleeplessness |
| | | Participant must score greater than or equal to a 5/10 for their primary symptom on the Baseline Symptom Questionnaire |
| | | Study cohort must have an available accrual slot for the participant respective of their primary symptom |
| | | Participant has signed the Informed Consent Form |

If any of the above boxes are checked "No", the subject does not meet eligibility criteria

Nu-V3 RCT PROTOCOL Eligibility Checklist V. 1.6 Version Date 21-Feb-2022



#### Nu-V3 RCT PROTOCOL

## EXCLUSION CRITERIA (all questions should be answered No – If question is answered Yes, subject is not eligible for participation)

| Yes | No | |
|---|---|---|
| | | Participants with a hearing aid |
| | | Participants with a pacemaker |
| | | Participants with an irregular heart rate or a heart rate lower than 60 beats per minute (bradycardia) |
| | | Have had a transplant within the last 2 years |
| | | Have had a heart attack or cardiac bypass surgery within the last 12 months |
| | | Patients with complaints of dizziness or lightheadedness within the last 3 months |
| | | Women who are pregnant |
| | | Participants with Diabetic Retinopathy |
| | | Current Ear infection |
| | | SBP < 100 and/or DBP < 60 |
| | | History of uncontrolled bipolar disorder within the last 12 months |
| | | History of uncontrolled seizures within the last 12 months |
| | | History of aneurysms |
| | | History of syncope within the last 12 months |
| | | Participants who have had a TIA or stroke within the last 12 months |
| | | Participants with health problems deemed at risk for the study by the Principal Investigator |
| | | Participants with any changes to Pain/Anxiety/Depression/Sleeplessness medications within last 60 days (participants that do not meet this medication change washout period may be delayed until 60-day period is met) |
| | | Participants that are currently under adjudication process for disability support, VA or other |

If any of the above boxes are checked "Yes", the subject does not meet eligibility criteria

Nu-V3 RCT PROTOCOL Eligibility Checklist V. 1.6 Version Date 21-Feb-2022


## **Appendix 3: IRB Unanticipated Problem Form**





| Nu-V3 Unanticipated Problem Form | | | | | | | |
|---|---|---|---|---|---|---|---|
| Nr. 372 | | | nitial Report: | | Follow-up No. | | Follow-up No. |
| Nu-V3<br>Version 1.0 | | | | | | | |
| Version Date:: 07/N | ov/2017 | - | id/mmm/yyyy | | dd / mmm / yyy | _ - | dd / mmm / yyyy |
| Investigator Name: | | | Site: | _ | da/mmi/yyy | Subject # | |
| | | | DEMO | GR | RAPHICS | , | |
| Gender | | | Date of Birth | Т | Height | | Weight |
| ☐ Female ☐ Male | | _ | /<br>dd / mmm / yyyy | | 🗆 in | □ cm | lbs |
| | | | | NT | INFORMAT | ION | |
| SAE Term (diagnosi | ADVERSE EVENT INFORMATION SAE Term (diagnosis preferred over signs/symptoms): | | | | | | |
| Onset Date | Grade | Outcome | | | | | |
| / / dd / mmm / yyyy Stop Date / / DD / MON / YYYY | hosp Life- Persi disab | italization<br>threaten<br>stent or<br>sility/inc<br>genital A<br>rtant me | | | Grade 1 - Mild Grade 2 - Mode Grade 3 - Seve Grade 4 - Life- Grade 5 - Fatal | rate<br>re<br>threatening | ☐ Ongoing ☐ Resolved ☐ Resolved w/ sequelae <sup>c</sup> ☐ Fatal |
| *Hospitalization: | Date | of Admi | ission / dd/mm | m/y | уууу р | ate of Discharg | e / / / dd / mmm / yyyy |
| Date of death | / /<br>l/mmm/ | уууу | Was autopsy complete<br>Is death certificate ava | | | | |
| Describe sequelae: | | | | | | | |
| | | | | | INFORMAT | | 1 10 11 |
| Study Device | | | Date of<br>First Use | | late of Last Use<br>efore SAE Onset | Relationship<br>to Device | Action taken<br>with Device |
| Nu-V3<br>□ N/A | _ | _ | | | / /<br>dd / mmm / yyyy | Related | ☐ None ☐ Dose Reduced ☐ Interrupted |
| Serial# | ther than | Study I | dd / mmm / yyyy | | | Unrelated | Discontinued |
| 1033DE CAUSE OF SAE O | _ | • | | | _ | Other, specif | r |
| | Con | dition to | Ma | dicat | ion name | | |

Document Title: Nu-V3 Unanticipated Problem Form

Effective Date: 07NOV2017 

| Nu-V3<br>Version 1.0<br>Version Date:: 07/Nov | /2017 | Site Na | me: | | | | Subject #: | | |
|---|---|---|---|---|---|---|---|---|---|
| Nu-V3 Treatment Modif<br>If action taken = interrupt<br>If action taken = interrupte | ed or discontinu | | • | | • | . – | Yes 🗌 No | | |
| RI | ELEVANT | LABOR | ATO | RY | DIAGNOS | STIC T | ESTS | None | |
| Test Name | | Dat<br>dd/mmm | | | Results/Va | due | Unit | | Normal Range |
| | | | | | | | | - | |
| | RELEVAN | T CONC | OM | TTA | NT MEDI | CATIO | NC D | <u> </u> | |
| | KELEVAN | CONC | OM | IIA | NI MEDI | Dose | ONS IN | one | |
| Medication | Start Date | | top D:<br>dd/m | ate or | Ongoing<br>7 | & Unit | Frequency | Route | Indication |
| | | | or | | oing | | | | |
| | | | or | _ | oing<br>oing | | | | |
| | | | or | _ | oing | | | | |
| | REL | EVANT | ME | DIC | AL HISTO | PRY | None | | • |
| Diagr | osis | | | | Start Date | | | | e or Ongoing |
| | | | | | drama yyyy | | | Ongoing | |
| | | | | | | | or | Ongoing | |
| | | | | | | | or | Ongoins | |
| | | NAI | RRA | TIV | E SUMMA | RY | | , ongoni | |
| Describe the even | nt in detail from o | onset throug | h reso | lution | . Include ration | nale for co | ausality and an | y interver | tions given. |
| | Describe the event in detail from onset through resolution. Include rationale for causality and any interventions given. | | | | | | | | |
| | | | RT | ER I | NFORMA | TION | | | |
| Investigator Name: | | Phone: | | | | | Email addre | 55: | |
| Reporter Name: Phone: Email address: | | | | | | | | | |
| INVESTIGATOR SIGNATU<br>L the | RE VERIFIES T | | | | | | | | |
| Signature: | | | | | Date: | | | | |
| Signature: | | | | | Date: | | | | |
| Signature: | Date: | | | | | | | | |

SAE report may be emailed to Nu-Life Solutions Executive Medical Team
Email: esiebeneck@nu-lifesolutions.com

Document Title: Nu-V3 Unanticipated Problem Form

Protocol Amendment 1.6 Date: 20-APR-2022

Effective Date: 07NOV2017 

## **Appendix 4: Adverse Event Form**

| Subject ID | _Date (dd/mmm/yyyy): | / | / |
|------------|----------------------|---|---|



#### **Adverse Events Form**

| 1. | Has the participant experienced any adverse events? |
|----|-----------------------------------------------------|
| | No (end of form)<br>Yes (update log below) |

#### 2. Adverse Event Log (CTCAE 5.0)

Grade 1=Mild Grade 2=Moderate Grade 3=Severe Grade 4=Life-threatening Grade 5=Death Attribution Grading: A=unrelated B=unlikely C=possibly D=probably E=definitely

| Event Name | SAE? | Grade | Attribution | Start Date<br>(dd/mmm/yyyy) | End Date<br>(dd/mmm/yyyy) | Treatment held or withdrawn? |
|---|---|---|---|---|---|---|
| | y/n | | ABCDE | | | |

Nu-Life Solutions Version Date: November 15, 2018

## **Appendix 5: Medical History Form**

| Subject ID | Date (dd/mmm/yyyy):/ |
|------------|----------------------|



#### Medical History Form

Please answer the following questions about your past and current medical history.

| 1. | o you have a history of any significant medical problems or chronic disease requiring a physician's care |
|---|---|
| | Yes (If Yes, please list below) 🔲 No |

| Medical Problem | Date of Diagnosis<br>(dd/mmm/yyyy) | Are you having trouble with this problem now? |
|---|---|---|
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |
| | / / | ☐ Yes ☐ No |

2. Have you had trouble with or sought medical attention for (please include even if stated in Question 1).

| Irregular Heart Rate | ☐ Yes ☐ No |
|----------------------|------------|
| Cardiac Arrhythmia | ☐ Yes ☐ No |
| Heart Disease | ☐ Yes ☐ No |

Nu-Life Solutions

| Subject ID | Date (dd/mmm/yyyy): | | |
|---|---|---|---|
| Chest Pain | □ Yes □ No | | |
| Heart Attack | ☐ Yes ☐ No | | |
| Heart Murmur | ☐ Yes ☐ No | | |
| Dizziness/ Lightheadedness | ☐ Yes ☐ No | | |
| Diabetic Retinopathy | ☐ Yes ☐ No | | |
| Bradycardia | ☐ Yes ☐ No | | |
| Epilepsy, Seizures, or Convulsions | ☐ Yes ☐ No | | |
| Aneurysms | ☐ Yes ☐ No | | |
| Syncope | ☐ Yes ☐ No | | |
| TIA or Stroke | ☐ Yes ☐ No | | |
| Drugs or Alcohol | ☐ Yes ☐ No | | |
| <ol> <li>Have you had trouble with or sought medic</li> </ol> | al attention for (please include ever | ı if stat | ed in Question 1). |
| High Blood Pressure | High Blood Pressure ☐ Yes ☐ No | | |
| Head Injury | ☐ Yes ☐ No | | |
| Chronic Neck or Back Pain | ☐ Yes ☐ No | | |
| Hypothyroidism | ☐ Yes ☐ No ☐ : | | ☐ Stable ☐ Unstable |
| Hyperthyroidism | ☐ Yes ☐ No | | Stable 🗆 Unstable |
| Rheumatoid Arthritis | ☐ Yes ☐ No | | |
| Inflammatory Arthritis | ☐ Yes ☐ No | | |
| Psoriatic Arthritis | ☐ Yes ☐ No | | |

Nu-Life Solutions

| Subject ID | Date (dd/mmm | /уууу): | <i></i> |
|---|---|---|---|
| Irritable Bowel Syndrome | ☐ Yes ☐ | No | |
| Neuropathy | ☐ Yes ☐ | No | ☐ Motor ☐ Sensory |
| Headaches | ☐ Yes ☐ I | No | ☐ Tension ☐ Migraine |
| 4. FEMALES ONLY; if male, skip to Question #5. a. Are you pregnant, or trying to become pregnant? Yes No b. Are you using birth control? Yes No c. If 'Yes', describe: 5. Have you had any surgery in the past three months? Yes No If 'Yes', describe: | | | |
| Depression | ☐ Yes ☐ No | □ 3-1 | s than 3 months ago<br>2 months ago<br>sater than 1 year ago |
| Bipolar Disorder | ☐ Yes ☐ No | Less than 3 months ago 3-12 months ago Greater than 1 year ago | |
| Panic Disorder | ☐ Yes ☐ No | □ 3-1 | s than 3 months ago<br>2 months ago<br>ater than 1 year ago |
| Phobia | ☐ Yes ☐ No | □ 3-1 | s than 3 months ago<br>2 months ago<br>eater than 1 year ago |

Nu-Life Solutions

| Subject ID | Date (dd/mmm, | /yyyy):/ |
|---|---|---|
| PTSD | ☐ Yes ☐ No | ☐ Less than 3 months ago ☐ 3-12 months ago ☐ Greater than 1 year ago |
| Obsessive Compulsive Disorder | ☐ Yes ☐ No | Less than 3 months ago 3-12 months ago Greater than 1 year ago |
| General Anxiety Disorder | ☐ Yes ☐ No | ☐ Less than 3 months ago ☐ 3-12 months ago ☐ Greater than 1 year ago |
| Schizophrenia | ☐ Yes ☐ No | Less than 3 months ago 3-12 months ago Greater than 1 year ago |
| Schizo-Affective Disorder | ☐ Yes ☐ No | Less than 3 months ago 3-12 months ago Greater than 1 year ago |
| 9. Have you ever been given any medications for emotional problems, such as anti-depressant, anti-anxiety or anti-psychotic medications? ☐ Yes ☐ No | | |

Nu-Life Solutions

## **Appendix 6: Treatment Form**



## **Weekly Treatment Form**

| Subject ID | Date (dd/mmm/yyyy):/ |
|-----------------------|------------------------------------|
| 1. Device Serial Numl | ber: |
| 2. Was the device pla | ced on the participant's left ear? |
| ☐ Yes ☐ No | If no, reason why: |

**Nu-Life Solutions** 

## **Appendix 7: Medications and Standard of Care Treatment Form**

| Subject ID | Date (DD/MMM/YYYY): | / | / |
|------------|---------------------|---|---|



#### **Medications and Standard of Care Treatment Form**

Please record all medications and other standard of care treatments related to any of the study indications, chronic pain, anxiety, depression, or sleeplessness. Include any treatments, supplements, and alternative holistic therapies.

| 1. Have the participant's medications changed? |
|---|
| No (continue to other treatments section) Yes (update the medications log below) |
| <ol> <li>Medications Log – Include any medications, herbal/non-herbal supplements, or<br/>medical marijuana used in the treatment of symptoms for chronic pain, anxiety,<br/>depression, or sleeplessness.</li> </ol> |

| Med Name | Dose | Unit | Frequency | Start Date<br>(dd/mmm/yyyy) | End Date<br>(dd/mmm/yyyy) | Indication |
|---|---|---|---|---|---|---|
| <u> </u> | | | | | | |

Nu-Life Solutions

Version Date: December 30, 2021

3. Treatment Log - Include any treatments related to symptom relief for chronic pain, anxiety, sleeplessness, or depression.

Examples include but are not limited to:

Aromatherapy
 Acupuncture

• Cryotherapy • Meditation

Tai Chi

| Start Date<br>(dd/mmm/yyyy) | End Date<br>(dd/mmm/yyyy) | Indication |
|---|---|---|
| | Start Date<br>(dd/mmm/yyyy) | Start Date (dd/mmm/yyyy) |

Nu-Life Solutions

Version Date: December 30, 2021

## **Appendix 8: ePRO Questionnaires**



| DATE: | Device/Pad serial # |
|--------|---------------------|
| Week # | Subject ID |

Complete Patient ePRO Questionnaire Packet



## Form DQ-7: Patient Demographics

| Subject ID | Race/Ethnicity |
|---|---|
| | Self-Description (please choose one): |
| | American Indian |
| Date (dd/mmm/yyyy): | Asian-American/Oriental/Pacific Islander |
| | Asian East Indian |
| | Black/African-American |
| Age | Mexican-America/Chicano |
| What is your age? | Puerto-Rican |
| | Other Hispanic |
| Sex at Birth | White/Caucasian |
| Male | Other |
| Female | |
| Other | Education History |
| Choose not to answer | What is the highest degree or level of school<br>you have completed? If currently enrolled, |
| | highest degree received. |
| Marital Status | No schooling completed |
| Single | Nursery school to 8th grade |
| Married | Some high school, no diploma |
| Divorced | High school graduate, diploma or GED |
| Widowed | Some college credit, no degree |
| P. ( | Trade/technical/vocational training |
| Primary Language? | Associate degree |
| Self-Description (please choose one): | Bachelor's degree |
| Arabic | Master's degree |
| Bengali | Professional degree |
| English<br>French | Doctorate degree |
| German<br>Hindi/Urdu | Service Status |
| Japanese | Are you now, or have you ever served as a |
| | member of the armed forces? |
| Portuguese | Yes, I am a military veteran |
| Portuguese<br>Punjabi | Yes, I am an active duty member |
| Russian | No, I have never served in the armed forces |
| Spanish | Are you a First Despendent Single-base Take In- |
| Other | Are you a First Responder (firefighter, EMS, law |
| | enforcement, etc)? |
| | Yes, I am current or former First Responder No, I have never been a First Responder |



## PEG: A Three-Item Scale Assessing Pain Intensity and Interference

| ubject ID: | | | | Date ( | dd/mm | m/yyyy | /): | / | _/_ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PEG: A | Thre | e-Item | Scale | Asses | s <b>ing</b> P | ain In | tensity | y and l | Interfe | erence | |
| 1. W | hat nu | mber b | est des | cribes y | your <u>pa</u> | in on a | verage | in the p | oast we | ek? | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| No pain | | | | | | | | | _ | Pain as ba<br>1 can ima | |
| | | mber b<br>r <u>enjoy</u> | | | how, du | ıring th | e past v | week, p | <b>ain ha</b> s | interfer | ed |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| No pain | | | | | | | | | | Pain as ba<br>1 can ima | |
| | | mber b<br>r gener | | | how, du | uring th | e past 1 | week, p | ain has | interfer | ed |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Pain as ba | 4 |
| No pain | | | | | | | | | | can ima | |

From Krebs et al., 2009.



#### GAD-7 - Generalized Anxiety Disorder 7-item Scale

| ld/mmm/yy | yy): | // | _ |
|---|---|---|---|
| Not at all sure | Several<br>days | Over half<br>the days | Nearly<br>every day |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| + | + | + | |
| | Not at all sure 0 0 0 0 0 0 0 | Not at all sure days 0 1 0 1 0 1 0 1 0 1 0 1 0 1 0 | all sure days the days 0 1 2 0 1 2 |

Source: Spitzer RL, Kroenke K, Williams JBW, Lowe B. A brief measure for assessing generalized anxiety disorder. Arch Inern Med. 2006;166:1092-1097.

care of things at home, or get along with other people?

Not difficult at all \_\_\_\_\_\_ Somewhat difficult \_\_\_\_\_

Extremely difficult \_\_\_\_\_

Very difficult \_\_\_

Protocol Amendment 1.6 Date: 20-APR-2022



## PHQ-9- Patient Health Questionnaire

| Subject ID: Date (d | d/mmm/yyy | /y <b>)</b> : | J | |
|---|---|---|---|---|
| Over the last 2 weeks, how often have you been | | | | |
| bothered by any of the following problems? (use "✓" to indicate your answer) | Not at all | Several<br>days | More than half the days | Nearly<br>every day |
| 1. Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| 2. Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| 3. Trouble falling or staying asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. Feeling tired or having little energy | 0 | 1 | 2 | 3 |
| 5. Poor appetite or overeating | 0 | 1 | 2 | 3 |
| Feeling bad about yourself—or that you are a failure or have let yourself or your family down | 0 | 1 | 2 | 3 |
| 7. Trouble concentrating on things, such as reading the<br>newspaper or watching television | 0 | 1 | 2 | 3 |
| 8. Moving or speaking so slowly that other people could<br>have noticed. Or the opposite — being so figety or<br>restless that you have been moving around a lot more<br>than usual | 0 | 1 | 2 | 3 |
| Thoughts that you would be better off dead, or of hurting yourself | 0 | 1 | 2 | 3 |
| | add columns | | + | + |
| (Healthcare professional: For interpretation of TOT please refer to accompanying scoring card). | AL, TOTAL: | | | |
| 10. If you checked off any problems, how difficult have these problems made it for you to do your work, take care of things at home, or get along with other people? | | | icult at all<br>hat difficult<br>ficult | |
| | | Extreme | ely difficult | |



## PROMIS Item Bank v1.0 - Sleep Disturbance - Short Form 4a

| Subject ID: | | Date (dd/i | mmm/yyyy) | :/_ | / | |
|---|---|---|---|---|---|---|
| | In the past 7 days | Very poor | Poor | Fair | Good | Very good |
| 1 | My sleep quality was | | | | | |
| | In the past 7 days | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| 2 | My sleep was refreshing. | | | | | |
| 3 | I had a problem with my sleep | | | | | |
| 4 | I had difficulty falling asleep | | | | | |



## PATIENTS' GLOBAL IMPRESSION OF CHANGE (PGIC) SCALE

| Subject ID: D | | | | (dd/mmm/yyyy) | | |
|---|---|---|---|---|---|---|
| Chief Complain | nt (Presenting | Problem): | | | | |
| LIMITATIONS, condition? Ple | SYMPTOMS ase circle the | , EMOTIONS, a | and OVERALL that matches | describe the conductive describe the conductive described the conductiv | LIFE, related | to your painful |
| No change | Almost the same | A little better | Somewhat better | Moderately better | Better | A great deal better |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Explanation: | | | | | | |
| 1 = No char | nge (or condition | has got worse) | 5 | = Moderately bet | ter, and a slig | ght but noticeable |
| 2 = Almost | the same, hardly | y any change at a | | change | | 197.10 |
| | | ticeable change | | <ul> <li>Better, and a def</li> <li>a real and worth</li> </ul> | | |
| | hat better, but the<br>difference | ne change has not | | = A great deal | better, and | |
| Patient's signa | ture: | | | | | |

#### NOTE TO HEALTH CARE PROVIDER

A significant, favorable change is a score of 5-7.

No significant change is a 1-4 response.

Note, this a dichotomous scale (5-7 = yes; 1-4 = no).

A 2-point change is significant from their last reported score.

Reference: Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. Journal of Manipulative Physiological Therapeutics (IMPT) 2004;27:26-35.

| Subject ID_ | Date (DD/MMM/YYYY): _ |
|-------------|-----------------------|



#### Form PTB-6: Patient's Perceived Treatment Benefit

 On a scale of 0-10, how much benefit do you feel you have received from the Nu-V3 treatment in helping your symptoms?



2. On a scale of 0-10, how much has your daily activity level improved?



3. Do you feel that your as needed medications have decreased from using the device?

\_\_\_\_Yes \_\_\_\_No

4. How comfortable was the Nu-V3 Device to wear?



5. Have you had any major discomfort from the device?

\_\_\_\_\_Yes; please continue to question 6
\_\_\_\_\_No

6. If yes to question 5, did adjusting the device correct the discomfort?

\_\_\_\_Yes No

Nu-Life Solutions

Version Date: March 2, 2022

## **Appendix 9: Baseline Symptom Questionnaire**



## **Baseline Symptom Questionnaire**

Please choose your primary symptom: (circle only one)

- rease anose your primary symptom (anote only one)
  - a. Chronic Pain b. A
- b. Anxiety
  - c. Depression
- d. Sleeplessness

Please rate your primary symptom over the last 30 days:

Pain Level:



Anxiety Level:



Depression Level:



Sleep Interruption Level:

